CLINICAL TRIAL: NCT03942432
Title: A Prospective, Mono-center, Interventional Study Evaluating the Effect of One Year Initial Care by Hygieno-dietary Advices With or Without Phlebotomy on Glycemia After at Least 5 Years in Patients With Dysmetabolic Iron Overload Syndrome
Acronym: EvoHSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC18_8847_EvoHSD
Record Dates: First submitted 2019-04-26; First posted 2019-05-08 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Dysmetabolic Iron Overload Syndrome
MeSH Terms: interventions — Glucose Tolerance Test; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with dysmetabolic iron overload syndrome (Experimental)
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Clinical exam; Biological: Blood sample; Device: MRI; Device: Bioimpedance; Behavioral: Questionnaires

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — Blood samples at T0, T30min, T120min
Other: Clinical exam — weight, length, waist measurement, cardiac frequency, blood pressure
Biological: Blood sample — Iron and cardiac markers Serum iron, serum transferrin, transferrin saturation, serum ferritin, AST, ALT, GGT, ALP, PT, Cell Blood Count, ceruloplasminemia , hyaluronic acid, cholesterolemia, HDL, LDL, triglyceridemia, hba1c
Device: MRI — 3 Tesla abdominal MRI
Device: Bioimpedance — Measurement of body composition
Behavioral: Questionnaires — Quality of life, physical activity, alcohol consumption and eating habits

SUMMARY:
A prospective, mono-center, interventional study evaluating the effect of one year initial care by hygieno-dietary advices with or without Phlebotomy on glycemia after at least 5 years in Patients with dysmetabolic iron overload syndrome

DETAILED DESCRIPTION:
Dysmetabolic iron overload syndrome (DIOS) is defined by a slight iron overload associated to features of the metabolic syndrome. This is a frequent condition that parallels the increasing prevalence of non alcoholic steato hepatitis. The role of iron overload on insulin sensitivity is described in large cohorts study, with an increased risk of type 2 diabetes in patients with increased serum ferritin, and in vitro where iron load alters key regulators of lipid and glucose metabolism.

In patient with DIOS, improving diet and lifestyle is a major goal, albeit it does not allow to lower body iron stores. Therefore the role of bloodletting in this setting was raised. Several low quality studies suggested a beneficial effect of bloodletting on insulin resistance. Our group demonstrated in a large multicenter randomized trial, the lack of beneficial effect of bloodletting over one year. Because this may be a too short period of time to demonstrate a positive effect we would like to assess the long term effect of iron depletion on insulin resistance and its clinical consequence.

ELIGIBILITY:
Inclusion Criteria:

* Persons who participated in the " Phlebotomy " protocol: A Prospective, Randomized Study Comparing Effect of Phlebotomy and Hygieno-dietary Advices With Hygieno-dietary Advices Only on Glycemia in Patients With Dysmetabolic Iron Overload Syndrome
* Persons affiliated to French Social Security
* Persons who received an oral and written information on the protocol and signed the informed consent form

Exclusion Criteria:

* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship) since their enrolment in the "Phlebotomy" protocol
* Persons deprived of liberty
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Dosage of fasting blood glycemia after 5 years | Year 5
  Oral Glucose Tolerance Test (OGTT)

SECONDARY OUTCOMES:
Dosage of iron hepatic concentration proved by MRI after 5 years | Year 5
  Abdominal MRI
Dosage of iron hepatic concentration after 5 years | Year 5
  Blood sample
Dosage of insulin after 5 years | Year 5
  Blood sample
Measurement of body composition | Year 5
  Bioimpedance
Measurement of insulin resistance markers | Year 5
  Oral Glucose Tolerance Test (OGTT)
Measurement of hepatic steatosis after 5 years | Year 5
  Abdominal MRI
Evaluation of cardiovascular morbi-mortality after 5 years | Year 5
  Mixed score based on the following events: angina pectoris, cardiac arrest, stoke
Calculation of Framingham score | Year 5
  Appreciation of cardiovascular event after 10 years based on blood pressure, cholesterol level and HDL, smoking or not, age and gender
Evaluation of quality of life after 5 years | Year 5
  SF-36 questionnaire
Evaluation of physical activity after 5 years | Year 5
  Baecke physical activity questionnaire : scores for physical exercise in leisure, leisure and locomotion activities
Evaluation of eating habits after 5 years | Year 5
  Eating habits questionnaire
Evaluation of alcohol consumption after 5 years | Year 5
  Alcohol consumption questionnaire : number of units of alcohol consumed per day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France